CLINICAL TRIAL: NCT06747546
Title: Research on Circulation Management Strategy Based on Oxygen Metabolism Balance After Congenital Heart Disease Surgery
Brief Title: Research on Circulation Management Strategy Based on Oxygen Metabolism Balance After CHD Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202501011231
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Congenital Heart Disease (CHD); Cardiopulmonary Bypass; Children; Oxygen Delivery; Oxygen Consumption; Oxygen Saturation; Goal-directed Therapy
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Treatment is routinely adjusted according to the changes of blood pressure and other monitoring indicators.Ventilation assistance is modified to sustain arterial oxygen partial pressure and oxygen saturation levels. Administer suitable fluid infusion to stabilize central venous pressure and maintain preload; Concurrent use of vasoactive agents to sustain heart rate and blood pressure; Effective diuresis can enhance urine production and decrease cardiac afterload. Blood transfusion is employed to enhance coagulation function and sustain adequate hematocrit levels.
  Interventions: Procedure: Conventional Treatment group
- Experimental group (Experimental): On the basis of routine treatment in the control group, PICCO is used to evaluate cardiac index (CI), bedside echocardiography is used to evaluate cardiac function, NIRS is used to measure rScO2, rSrO2 and rSsO2, and arterial and central venous blood gas are measured at the same time after operation. DO2, VO2, ERO2, and Pv-aCO2 gap are calculated according to the formula. The oxygen extraction rate immediately after CPB is set as E1, the oxygen extraction rate at 4 hours after surgery is E2, and the oxygen extraction rate at 8 hours after surgery is E3.A "goal-directed" treatment strategy based on oxygen supply and consumption balance is defined as: Combined with the value of E2 at 4 hours after CPB, the increasing VO2 after CPB is compensated by increasing DO2 to different degrees. The goal of E3 not increasing significantly compared with E1 is achieved at 8 hours after CPB, and the severity of low cardiac output is finally reduced within the "golden 8 hours" after CPB.
  Interventions: Procedure: "goal-directed" treatment strategy based on oxygen supply and consumption balance

INTERVENTIONS:
Procedure: "goal-directed" treatment strategy based on oxygen supply and consumption balance — The oxygen extraction rate immediately after CPB is set as E1, the oxygen extraction rate at 4 hours after surgery is E2, and the oxygen extraction rate at 8 hours after surgery is E3. A "goal-directed" treatment strategy based on oxygen supply and consumption balance is defined as: Combined with the value of E2 at 4 hours after CPB, the increasing oxygen consumption (VO2) after CPB is compensated by increasing oxygen delivery (DO2) to different degrees. The goal of E3 not increasing significantly compared with E1 is achieved at 8 hours after CPB, and the severity of low cardiac output is finally reduced within the "golden 8 hours" after CPB.
  Arms: Experimental group
Procedure: Conventional Treatment group — Ventilation support is adjusted to maintain arterial oxygen partial pressure and oxygen saturation. Appropriate fluid infusion to stabilize central venous pressure and ensure preload; Combined use of vasoactive drugs to maintain heart rate and blood pressure; Appropriate diuresis can improve urine output and reduce cardiac afterload. Blood transfusion is used to improve coagulation function and maintain appropriate hematocrit.
  Arms: Control group

SUMMARY:
The objective is to investigate a goal-oriented postoperative circulation management strategy centered on "oxygen metabolism balance". This strategy is independent of the absolute metrics of oxygen supply and consumption, and aims to enhance oxygen consumption and uptake within the critical "golden 8 hours" following pediatric cardiopulmonary bypass, thereby preventing severe hypotension, cardiopulmonary arrest, and other adverse events.

DETAILED DESCRIPTION:
This study firstly offered a specialized treatment strategy for children, particularly those who have undergone cardiopulmonary bypass surgery, that uses tailored parallel control and is independent of absolute oxygen supply and consumption characteristics.In addition, this study seeks to investigate the correlation between oxygen supply and consumption following pediatric cardiopulmonary bypass surgery and to assess the clinical utility of a goal-directed strategy concerning cardiac function recovery (ICON, echocardiography, myocardial markers) and outcomes (incidence of low cardiac output, duration of endotracheal intubation, length of CCU stay, and mortality). This strategy is of great significance to improve the surgical outcomes and prognoses for children.

ELIGIBILITY:
Inclusion Criteria:

* 1.Body weight > 2.5kg;
* 2.Preoperative oxygen saturation >80%;
* 3.Biventricular radical surgery with cardiopulmonary bypass.

Exclusion Criteria:

* 1. Complicated with functional single ventricle and atrial isomerism;
* 2.Complicated with liver, kidney, lung, brain and other vital organ diseases;
* 3.History of rescue before operation;
* 4.Palliative surgery;
* 5.Residual deformities that significantly affected hemodynamics after operation;
* 6.Guardians did not provide the bundle of informed consent.

Ages: 1 Week to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 300 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with low cardiac output syndrome | 72 hours after surgery
  Low Cardiac Output Syndrome (LCOS) is a pathological state of cardiac dysfunction, which is usually manifested as a significant decrease in cardiac output (the amount of blood pumped by the heart per minute), leading to hypoperfusion of systemic organs.Low cardiac output was defined as cardiac index <2.0L/(min.m2).

SECONDARY OUTCOMES:
Number of death | 1 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ping Ya Mi, Study Director — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Minhang, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No